CLINICAL TRIAL: NCT01561417
Title: A Single-centre, Randomised, Double-blind, Two-way Cross-over Trial Investigating the Bio-equivalence in Healthy Male Subjects of NovoSeven (CP-rFVIIa) and a Formulation of NovoSeven Stable at 25°C (VII25)
Brief Title: Bioequivalence of NovoSeven® and a NovoSeven® Formulation Stable at Room Temperature in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN1007-1744; 2005-005379-14 (EudraCT Number)
Record Dates: First submitted 2012-03-21; First posted 2012-03-23 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Acquired Bleeding Disorder; Acquired Haemophilia; Congenital Bleeding Disorder; Congenital FVII Deficiency; Glanzmann's Disease; Haemophilia A With Inhibitors; Haemophilia B With Inhibitors; Healthy
MeSH Terms: conditions — Thrombasthenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CP-rFVIIa (Active Comparator)
  Interventions: Drug: activated recombinant human factor VII
- VII25 (Experimental)
  Interventions: Drug: activated recombinant human factor VII

INTERVENTIONS:
Drug: activated recombinant human factor VII — One single dose administration, injected i.v. (into the vein)
  Arms: CP-rFVIIa
Drug: activated recombinant human factor VII — One single dose administration, injected i.v. (into the vein)
  Arms: VII25

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to demonstrate bio-equivalence between the marketed activated recombinant human factor VII (NovoSeven®) (CP-rFVIIa) and a new formulation stable at 25°C (VII25).

ELIGIBILITY:
Inclusion Criteria:

* Caucasian
* Body Mass Index (BMI) between 18 and 27 kg/m^2, both inclusive
* Good health as indicated by medical history, physical examination including vital signs and ECG, and clinical laboratory test results
* Smoke less than 10 cigarettes (or equivalent) per day
* Capable of giving written Informed Consent (IC)

Exclusion Criteria:

* Evidence of clinically relevant pathology or potential thromboembolic risk based on medical and/or family history as judged by the Investigator
* Known history of atherosclerosis, arteriosclerosis, thromboembolic events or known high levels of Troponin I
* Known or suspected allergy to activated recombinant human factor VII or related products or any of the components of the formulation
* Overt bleeding, including from gastrointestinal tract
* Hepatitis (B or C) infection
* HIV (human immunodeficiency virus) infection

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2006-04; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve for FVIIa clot activity

SECONDARY OUTCOMES:
The maximum plasma concentration (Cmax)
Terminal half-life (t½)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Paris, France

REFERENCES:
- [Result] Bysted BV, Scharling B, Moller T, Hansen BL. A randomized, double-blind trial demonstrating bioequivalence of the current recombinant activated factor VII formulation and a new robust 25 degrees C stable formulation. Haemophilia. 2007 Sep;13(5):527-32. doi: 10.1111/j.1365-2516.2007.01516.x. PMID 17880439
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com